CLINICAL TRIAL: NCT07226557
Title: Cefiderocol vs Best Available Therapy for Carbapenem-resistant Acinetobacter Baumannii-calcoaceticus Complex Infections: A Target Trial Emulation
Status: Active, not recruiting | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: BD070725
Record Dates: First submitted 2025-11-05; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-07

CONDITIONS: Carbapenem Resistant Bacterial Infection; Acinetobacter Baumannii Infection; Antimicrobial Drug Resistance
Keywords: Carbapenem-resistant Acinetobacter baumannii; Cefiderocol; Target trial emulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reciept of cefiderocol: Inpatients with carbapenem-resistant Acinetobacter baumannii infection that receive empiric and/or targeted therapy including cefiderocol.
- Reciept of best available therapy (BAT): Inpatients with carbapenem-resistant Acinetobacter baumannii infection that receive empiric and/or targeted therapy with activity against the infection but does not include cefiderocol

SUMMARY:
This study aims to compare 28-day mortality among patients with carbapenem resistant A. baumannii infections in two hypothetical target trials where patients receive 7 days of a cefiderocol-based treatment strategy or 7 days of a best available therapy treatment strategy.

DETAILED DESCRIPTION:
please see uploaded study protocol

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adults (≥ 18 years of age)
* Carbapenem resistant A. baumannii-calcoaceticus complex clinical culture
* Antimicrobial agent with possible in vitro activity against carbapenem resistant A. baumannii-calcoaceticus complex initiated in the time frame of 2 days before culture collection until 2 days following first available antibiotic susceptibility test result being made available

Exclusion Criteria:

* Patients with no antibiotic susceptibility testing
* Patients with only A. baumannii infection diagnosed by rapid diagnostic tests (i.e., multiplex polymerase chain reaction)
* Initiation of antimicrobial agent outside of selected time frame (i.e., 2 days before culture collection until 2 days after first available antibiotic susceptibility test result was made available)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized adult patients with a clinical culture positive for carbapenem resistant A. baumannii and received an antibiotic with possible in vitro activity against carbapenem resistant A. baumannii in the time frame of interest (i.e., days before culture collection until 2 days after first available antibiotic susceptibility test result was made available) and admitted to US hospitals reporting to the PINC-AI healthcare database between 2018-2024 will be eligible for inclusion in the hypothetical target trials.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | During inpatient admission
  In hospital mortality or discharge to hospice during the hospital stay

SECONDARY OUTCOMES:
Length of Stay | Inpatient admission
  Duration of hospitalization among surviving patients
Recurrent CRAB Infection | Within 30 days post discharge
  clinical culture positive for carbapenem-resistant A. baumannii (CRAB) infection within the same encounter downstream of the index episode and within 30 days.
Development of antibiotic resistance to initial antibiotic treatment | Subsequent admissions
  Development of antibiotic resistance on a subsequent positive clinical culture to an antibiotic administered during prior infectious episode

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Kadri, MD, Principal Investigator — National Institutes of Health CC
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data, analytic methods, and data dictionary will be shared upon request to the primary contact.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT07226557/Prot_SAP_000.pdf